CLINICAL TRIAL: NCT03390972
Title: Effects of Dexmedetomidine on Swallowing Function: a Randomized, Double-Blind Study in Healthy Volunteers
Brief Title: Dexmedetomidine and Swallowing Function
Acronym: DexSwallow
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Region Örebro County (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: JS007
Record Dates: First submitted 2017-12-14; First posted 2018-01-05 (Actual); Last update posted 2018-01-05 (Actual); Status verified 2017-12

CONDITIONS: Deglutition
Keywords: Dexmedetomidine; Swallowing function; Anesthetic sedation
MeSH Terms: interventions — Sodium Chloride; Dexmedetomidine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dexmedetomidine (Experimental): Volunteers are given an intravenous infusion with dexmedetomidine, with an effect-site target concentration of 0.6 ng/ml via a target-controlled infusion (TCI) pump. After a series of swallowing tests the effect-site target concentration is raised to 1.2 ng/ml and the swallowing series is repeated.
  Interventions: Drug: Dexmedetomidine
- Placebo (Placebo Comparator): Volunteers are given an intravenous infusion with saline 0,9% with target controlled infusion pump in corresponding doses as in the dexmedetomidine arm.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Placebo — Placebo (NaCl 0.9%) TCI infusion
  Other Names: Sodium Chloride 0.9%
  Arms: Placebo
Drug: Dexmedetomidine — Dexmedetomidine TCI 0.6 ng/ml and 1.2 ng/ml
  Other Names: Dexdor
  Arms: Dexmedetomidine

SUMMARY:
The purpose of the study is to evaluate the impact of dexmedetomidine on swallowing function in healthy volunteers using combined pressure and impedance recordings. Furthermore, two different concentrations of dexmedetomidine will be studied to find out whether any posible impact of dexmedetomidine on swallowing function is dose-dependent.

DETAILED DESCRIPTION:
Monitored anesthesia care (MAC) is commonly applied in modern perioperative care and means that minor surgical procedures are accomplished in awake patients using local anesthesia and light sedation. MAC has many advantages compared to general anesthesia; the recovery time after anesthesia is shorter and risk for postoperative nausea is lower to mention some. However, the patient is spontaneously breathing and the airway is not protected by an endotracheal tube which potentially increases risk of pulmonary aspiration. Pulmonary aspiration, that is inhalation of stomach and/or pharyngeal contents into the lungs, is a severe anesthesia-related complication and can in worst case lead to pneumonia and even death. Intact swallowing function is crucial in avoiding aspiration and how sedatives and analgesic agents used during MAC influence swallowing function is not fully understood.

Pharyngeal function during bolus swallowing is measured by combined high resolution impedance manometry (HRIM). The HRIM catheter is inserted through the nose in such a way that sensors straddle the entire pharynx and esophagus with the distal catheter tip in the stomach. Dynamic pressure changes and flow can be detected during swallowing and data registered by HRIM are analysed using purpose-designed software, AIM analysis (automated impedance manometry analysis). AIM analysis derives pressure flow variables which describe different physiological events like bolus timing and bolus distension in the pharynx and the esophagus during swallowing. A Swallow Risk Index value, quantifying risk of deglutitive aspiration, can also be defined.

The aim of the study is to evaluate impact of dexmedetomidine on swallowing function in healthy volunteers.Dexmedetomidine is a selective alfa-agonist frequently used during MAC. Furthermore, two different concentrations of dexmedetomidine will be studied to find out whether any posible impact of dexmedetomidine on swallowing function is dose-dependent. Moreover, subjective swallowing difficulties will be assessed.

20 healthy volunteers will be studied on two different occasions approximately one week apart. In a randomized order volunteers will receive intravenous infusion of dexmedetomidine in two subsequent concentrations and placebo (normal saline) infusion in corresponding doses on the other occasion. Blood samples are obtained for plasma concentration determination of the study drug and sedation levels are assessed during study drug exposure.

ELIGIBILITY:
Inclusion Criteria:

1. ≥ 18 - ≤ 40 year old healthy volunteers from both sexes.
2. Have signed and dated Informed Consent.
3. Willing and able to comply with the protocol for the duration of the trial.

Exclusion Criteria:

1. Anamnesis of pharyngoesophageal dysfunction.
2. Known or history of gastrointestinal, severe cardiac, pulmonary or neurological disease
3. Ongoing medication that may affect upper gastrointestinal tract, larynx or lower airway.
4. Allergies to or history of reaction to remifentanil, fentanyl analogues or dexmedetomidine.
5. Known heart rhythm disorder.
6. Tendency to faint.
7. Pregnancy or breast feeding
8. BMI > 30
9. Smoking
10. Participation in a medicinal clinical trial during the last year where an opioid has been used or have during the last 30 days participated in any other medicinal clinical trial or in a trial where follow-up is not completed.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2018-01-22 (Estimated); Primary Completion 2018-04-11 (Estimated); Study Completion 2018-04-11 (Estimated)

PRIMARY OUTCOMES:
Swallow Risk Index, dex vs baseline | 60 minutes
  Global measure of swallowing dysfunction related to aspiration risk, during swallowing between dexmedetomidine exposure and baseline compared to placebo.
Hypopharyngeal Intrabolus Pressure, dex vs baseline | 60 min
  Measure of pharyngeal outflow resistance, mmHg
Mean Distension Contraction Latency, dex vs baseline | 60 min
  Measure of flow timing, sec
Hypopharyngeal Bolus Presence Time, dex vs baseline | 60 min
  Measure of bolus arrival/oral bolus control, sec
Velopharyngeal to Tongue Base Pressure Integral, dex vs baseline | 60 min
  Measure of lumen occlusive pressure, mmHgxsxcm
Hypopharyngeal Contractile Integral, dex vs baseline | 60 min
  Measure of lumen occlusive pressure, mmHgxsxcm
Mean Pharyngeal Peak Pressure, dex vs baseline | 60 min
  Measure of lumen occlusive pressure, mmHg
Mean UES Basal Pressure, dex vs baseline | 60 min
  Measure of UES (upper esophageal sphincter) basal tone, mmHg
UES Open Time, dex vs baseline | 60 min
  Measure of UES opening, sec
UES Maximum Admittance | 60 min
  Measure of UES opening, ms
UES Integrated Relaxation Pressure | 60 min
  Measure of UES relaxation, mmHg

SECONDARY OUTCOMES:
Pharyngeal Pressure Flow variables, dex 0.6 ng/ml vs 1.2 ng/ml | 60 minutes
  Difference in pressure flow variables during swallowing between dexmedetomidine target concentration of 0.6 ng/ml and 1.2 ng/ml compared to placebo.
Esophageal pressure flow variables, dex vs baseline | 60 min
  Difference in pressure flow variables during swallowing between dexmedetomidine exposure and baseline compared to placebo.
Esophageal pressure flow variables, dex 0.6 ng/ml vs 1.2 ng/ml | 60 min
  Difference in esophageal pressure flow variables during swallowing between dexmedetomidine target concentration of 0.6 ng/ml and 1.2 ng/ml compared to placebo.
Subjective swallowing difficulties | 60 minutes
  Difference in subjective swallowing difficulties between dexmedetomidine exposure and baseline compared to placebo.

CONTACTS AND LOCATIONS:
Overall Officials: Johanan Savilampi, Phd, Principal Investigator — Department of Anaesthesiology and Intensive Care, Örebro University Hospital

IPD SHARING:
Plan to Share IPD: No